CLINICAL TRIAL: NCT02721017
Title: Pain Control in the Nuss Procedure: A Prospective, Randomized Trial of Cryoanalgesia vs. Thoracic Epidural
Brief Title: Cryoanalgesia vs. Epidural in the Nuss Procedure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-18202; 1R03HD090617-01 (NIH); 1P50FD006424-01 (FDA)
Record Dates: First submitted 2016-03-22; First posted 2016-03-28 (Estimated); Results first posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Pectus Excavatum; Funnel Chest
Keywords: Nuss; Nuss Procedure; pectus excavatum; cryoanalgesia
MeSH Terms: conditions — Funnel Chest | interventions — Tea; Fentanyl; Injections, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Cryoanalgesia (Experimental): Cryoanalgesia performed thoracoscopically under general anesthesia by the patient's surgeon at the time of the Nuss procedure
  Interventions: Device: Cryoanalgesia
- Thoracic Epidural (Active Comparator): Thoracic epidural (ropivicaine, fentanyl).
  Interventions: Drug: Thoracic epidural (ropivicaine, fentanyl)

INTERVENTIONS:
Device: Cryoanalgesia
  Other Names: AtriCure; cryoprobe; nerve freezing
  Arms: Cryoanalgesia
Drug: Thoracic epidural (ropivicaine, fentanyl) — Epidural infusion was begun with with 0.1% ropivicaine and 2 mg/cc fentanyl.
  Other Names: Epidural
  Arms: Thoracic Epidural

SUMMARY:
The purpose of this study is to determine whether cryoanalgesia provides better pain control for minimally invasive pectus excavatum repair (the Nuss procedure) than thoracic epidural.

DETAILED DESCRIPTION:
Pain control is a major challenge for physicians, who must ensure appropriate and effective pain control for their patients, while remaining mindful of the many negative effects of opioid dependence and addiction. Nowhere is there a more pressing need than in children and young adults, who are at high risk for drug abuse, and in post-operative care, since post-operative opioid use can be a starting point for long-term pain issues. Postoperative pain control in the Nuss procedure, minimally invasive repair of the congenital chest wall deformity known as pectus excavatum, remains a significant problem for the 3000 patients who undergo this procedure each year, mostly adolescents and young adults. Many multimodal analgesic regimens have been tried, but optimal treatment remains unknown.

This study will test a novel and promising strategy of using intra-operative cryoanalgesia during the Nuss procedure. Cryoanalgesia is the localized, temporary freezing of peripheral nerves, which is performed at the time of the Nuss procedure. The study is a 20-subject prospective, randomized pilot trial comparing cryoanalgesia to thoracic epidural analgesia for post-operative pain control in patients undergoing the Nuss procedure. Subjects will be recruited from patients already scheduled for a Nuss procedure at our institution, and will undergo 1:1 randomization to either cryoanalgesia or thoracic epidural analgesia for perioperative pain control. During their hospitalization, patients' opiate usage will be prospectively recorded, and pain will be assessed twice per day. Upon discharge, patients will maintain a log of their opiate use, and will return to clinic at 2 weeks, 1 month, 3 months, and 1 year after Nuss procedure for post-operative assessment. Primary outcome is length of perioperative hospitalization, an objective measure that synthesizes many different aspects of a procedure and its subsequent post-operative course, including pain control. Secondary outcomes are post-operative narcotic usage and direct cost of perioperative hospitalization. Side effects of both interventions will also be assessed.

This will be the first systematic investigation of cryoanalgesia for local nerve block in a thoracoscopic procedure, and the first study involving its use in adolescents and young adults. The results will have direct application for those undergoing the Nuss procedure to repair pectus excavatum. Investigators will also delineate a reproducible protocol for delivering cryoanalgesia thoracoscopically, to ensure others can safely and effectively use this method if it proves beneficial. Although the focus is on the small subset of patients who undergo the Nuss procedure, if a standardized approach to cryoanalgesia delivery in a thoracoscopic procedure has a positive effect on patient outcomes and cost of hospitalization, the technique could be applied to a variety of surgical procedures, as well as for other neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for Nuss procedure for pectus excavatum correction
* at least 13 years old at the time of the procedure

Exclusion Criteria:

* age less than 13 years at time of procedure
* use of pain medication prior to procedure
* pectus carinatum, Poland's syndrome, or any chest wall anomaly other than pectus excavatum
* previous repair of pectus excavatum by any technique
* previous thoracic surgery
* congenital heart disease
* bleeding dyscrasia
* major anesthetic risk factors or history of previous problem with anesthesia
* pregnancy
* inability to communicate in English

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Padilla, MD, Principal Investigator — 415-370-2835
Locations (1):
- UCSF-Benioff Children's Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Graves C, Idowu O, Lee S, Padilla B, Kim S. Intraoperative cryoanalgesia for managing pain after the Nuss procedure. J Pediatr Surg. 2017 Jun;52(6):920-924. doi: 10.1016/j.jpedsurg.2017.03.006. Epub 2017 Mar 16. PMID 28341230
- [Result] Graves CE, Moyer J, Zobel MJ, Mora R, Smith D, O'Day M, Padilla BE. Intraoperative intercostal nerve cryoablation During the Nuss procedure reduces length of stay and opioid requirement: A randomized clinical trial. J Pediatr Surg. 2019 Nov;54(11):2250-2256. doi: 10.1016/j.jpedsurg.2019.02.057. Epub 2019 Mar 17. PMID 30935731

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty consecutive patients were recruited from those scheduled for the Nuss procedure.
Pre-assignment Details: Exclusion criteria were age <13 years, chest wall anomaly other than pectus excavatum, previous repair or other thoracic surgery, and chronic use of pain medications.
Groups:
- Cryoanalgesia: Cryoanalgesia performed thoracoscopically under general anesthesia by the patient's surgeon at the time of the Nuss procedure
  Cryoanalgesia
Period: Hospital Stay
Arm/Group | Cryoanalgesia | Thoracic Epidural
Started | 10 (Intraoperative Application of Cryoanalgesia started on Date of Surgery (DOS).) | 10 (Thoracic Epidural placed on Date of Surgery (DOS).)
Completed | 10 (Completed during the course of surgery.) | 10 (Removal occurs prior to Hospital Discharge.)
Not Completed | 0 | 0
Period: Participant Follow Up
Arm/Group | Cryoanalgesia | Thoracic Epidural
Started | 10 (Assessment of recovery at 2 weeks, 1 month, 3 month and 12 month intervals.) | 10 (Assessment of recovery at 2 weeks, 1 month, 3 month and 12 month intervals.)
Completed | 10 (12 months after Date of Surgery.) | 10 (12 months after Date of Surgery.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cryoanalgesia | Thoracic Epidural | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 7 | 11
  Between 18 and 65 years | 6 | 3 | 9
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 20.9 [14 to 31] | 16.1 [13 to 21] | 18.5 [13 to 31]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 9 | 8 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Length of Hospitalization
Description: the length of the patient's in-hospital stay following admission for Nuss procedure
Time Frame: estimated one week or less
Measure: Median (Full Range); unit: Length of Stay (Post-Operative Days)
Arm/Group | Cryoanalgesia | Thoracic Epidural
Number analyzed (Participants) | 10 | 10
Length of Stay (Post-Operative Days) | 3 [2 to 4] | 5 [4 to 6]

2. Secondary Outcome: Narcotic Usage
Description: Inpatient narcotic usage
Time Frame: Post Operative Hospital Stay
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Cryoanalgesia | Thoracic Epidural
Number analyzed (Participants) | 10 | 10
mg | 268 (165.2) | 684 (191.8)

3. Secondary Outcome: Mean Neuropathic Pain Score at One Year
Description: Neuropathic specific pain (described as "burning", "electrical" or "tingling" sensations) was assessed by study questionnaire via numerical pain scale (1 to 10, with 10 representing a maximum score, or worst pain possible).
Time Frame: one year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cryoanalgesia | Thoracic Epidural
Number analyzed (Participants) | 10 | 10
score on a scale | 2.4 (2.69) | 1.9 (1.34)

4. Secondary Outcome: Cost Analysis
Description: cost analysis of initial hospitalization following Nuss procedure
Time Frame: estimated one week
Population: Cost analysis was not performed, as these data were not collected.
Arm/Group | Cryoanalgesia | Thoracic Epidural
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: All adverse events reported post operatively at the 2 week, 1 month, 3 month and 1 year follow up points were collected. In addition all serious adverse events that occurred following enrollment were as well collected. The collection period for all serious adverse events began after informed consent was obtained and ended after procedures for the final study visit had been completed at the 1 year post-operative mark.
Arm/Group | Cryoanalgesia | Thoracic Epidural
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 2/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cryoanalgesia (N=10) | Thoracic Epidural (N=10)
Paraplegia (Nervous system disorders) | 0 (0) | 0 (0)
Symptomatic Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 0 (0) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Infection from indwelling thoracic epidural catheter (Infections and infestations) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-07): https://cdn.clinicaltrials.gov/large-docs/17/NCT02721017/Prot_SAP_000.pdf